CLINICAL TRIAL: NCT00834925
Title: Low Dose of Diltiazem for Rate Control of Atrial Fibrillation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Min Seung Chun, Mitsubishi-Tanabe Coperation Group
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Diltiazem Af
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation with rapid ventricular response
MeSH Terms: conditions — Atrial Fibrillation | interventions — Diltiazem

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- standard dose diltiazem (No Intervention)
- low dose diltiazem (Experimental)
  Interventions: Drug: low dose diltiazem

INTERVENTIONS:
Drug: low dose diltiazem — Low dose diltiazem: 0.15mg/kg over 2 minutes Standard dose diltiazem: 0.25mg/kg over 2 minutes
  Arms: low dose diltiazem

SUMMARY:
This study is to show the efficacy and safety of low dose diltiazem for the treatment of atrial fibrillation with rapid ventricular response in emergency room. We will compare the standard dose of diltiazem(0.25mg/kg) with low dose diltiazem(0.1mg/kg)in atrial fibrillation with rapid ventricular response in ED.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation with rapid ventricular response in emergency room

Exclusion Criteria:

* age<18
* systolic blood pressure<90mmHg
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Success rate of rate control | in 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea